CLINICAL TRIAL: NCT04382820
Title: Psychosocial Situation of Children With Rare (Congenital) Pediatric Surgical Diseases and Their Families
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Johannes Boettcher, Principial investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: PV7161
Record Dates: First submitted 2020-05-04; First posted 2020-05-11 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Rare Diseases
Keywords: rare diseases; pediatric surgery; children and adolescent; quality of life; psychological distress
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Families of rare chronically ill children: Clinical study participants for the diagnostic study are patients who have sought treatment at the University Medical Center Hamburg-Eppendorf due to a rare pediatric surgical disease. Every family receives a comprehensive psychosocial diagnostic in the form of standardized instruments.
- Families in the comparative control group: Participants in the healthy control sample are matched to the clinical sample in terms of age and gender. Included are families of children aged 0-21 years, who have undergone a surgical procedure in the first 3 years of life that does not cause chronic complaints; such as hernia surgery or testicular relocation.

SUMMARY:
Families of children with rare diseases (i.e., not more than 5 out of 10.000 people are affected) are often highly burdened with fears, insecurities and concerns regarding the affected child and his/her siblings. The aim of the present research project is to examine the psychosocial burden of the children with rare (congenital) pediatric surgical diseases and their family in order to draw attention to a possible psychosocial care gap in this population.

DETAILED DESCRIPTION:
The central objective of the cross-sectional study is to show the psychosocial supply gap for families with children and adolescents affected by rare diseases in the field of pediatric surgery. Among the rare diseases that are included are diaphragmatic hernia, anorectal malformations, esophageal atresia, Hirschsprung's disease and biliary atresia. In order to have a comparative sample, additional data of a matched control group are collected. Central standardized psychosocial outcomes will be assessed from the perspectives of the parents, the affected child and the siblings.

ELIGIBILITY:
Inclusion Criteria (families of rare disease):

* Family with at least one child between 0 and 21 years with a rare pediatric surgical disease.
* Consent to participate in the study.
* Sufficient knowledge of the German language of parents and children.

Exclusion Criteria (families of rare disease):

* Severe acute physical, mental and/or cognitive impairment of the child, so that the questionnaire survey does not appear possible and/or unreasonable at this stage.

Inclusion Criteria (control group):

* Family with at least one child between 0 and 21 years who have undergone a surgical procedure in the first 3 years of life that does not cause chronic complaints
* Consent to participate in the study.
* Sufficient knowledge of the German language of parents and children.

Exclusion Criteria (control group):

- Families of children with a congenital or chronic disease.

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Clinical study participants for the diagnostic study are patients who have sought treatment at the University Medical Center Hamburg-Eppendorf due to a rare pediatric surgical disease. Participants in the healthy control sample are matched to the clinical sample in terms of age and gender. Included are families of children aged 0-21 years, who have undergone a surgical procedure at the University Medical Center Hamburg-Eppendorfin the first 3 years of life that does not cause chronic complaints; such as hernia surgery or testicular relocation.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Quality of life of the parents (ULQIE) | 4 minutes
  Quality of life (QoL) of the parents, assessed from the perspective of the parents by the "Ulmer Lebensqualitätsinventar für Eltern chronisch kranker Kinder" (ULQIE; Goldbeck & Storck, 2002). The instrument consists of 29 items, which are answered on a five-point Likert scale (0 to 4). Higher scores indicate greater QoL.
Mental health of the parents (BSI) | 5 minutes
  Mental health of the parents, assessed from the perspective of the parents by the "Brief Symptom Inventory" (BSI; Franke, 2000). The instrument consists of 53 items, which are answered on a five-point Likert scale (0 to 4). Higher BSI scores indicate greater psychological distress.
Health-related quality of life of the chronically-ill children/adolescents (Peds-QL 4.0) | 4 minutes
  Health-related quality of life of the chronically-ill children/adolescents, assessed from the perspective of the child/adolescent (from 10 years of age) and from the perspective of the parents by the "Pediatric Quality of Life Inventory 4.0" (Peds-QL 4.0; (Varni, Seid, & Kurtin, 2001). Items will be linearly transformed to a scale of 0 to 100, with higher scores indicating better HRQoL.
Psychiatric disorders of the chronically-ill children/adolescents and the siblings (SDQ) | 4 minutes
  Psychiatric disorders of the chronically-ill children/adolescents and the siblings assessed perspective of the child/adolescent (from 10 years of age) and from the perspective of the parents by the "Strengths and Difficulties Questionnaire" (SDQ; Klasen, Woerner, Rothenberger, & Goodman, 2003). Items are rated on a three-point Likert scale (0 to 2). Higher scores represent greater psychopathology or greater prosocial behavior.

SECONDARY OUTCOMES:
Coping of the parents (CHIP-D) | 3 minutes
  Coping of the parents, assessed from the perspective of the parents by the German version of the "Coping Health Inventory for Parents" (CHIP-D; McCubbin, McCubbin, Cauble & Goldbeck, 2001). Items are rated on a four-point Likert scale (0 to 3). Higher scores represent greater use of the respective coping pattern.
Coping of the chronically-ill children/adolescents and the siblings (Kidcope) | 3 minutes
  Coping of the chronically-ill children/adolescents and the siblings, assessed from the perspective of the children/adolescents (from 10 years of age) by the "Kidcope Checklist" (Kidcope; Spirito, Stark & Williams, 1988). Items related to frequency of the coping strategies are rated on a 4 point scale (0 = "Not at all" to 3 = "Almost all the time"), and items related to efficacy are rated on a 5 point scale (0 = "Not at all" to 4 = "Very much").
Social support of the parents, of the chronically-ill children/adolescents and of the siblings (OSSS) | 3 minutes
  Social support of the parents, of the chronically-ill children/adolescents and of the siblings, assessed from the perspective of the parents, of the chronically-ill children/adolescents and from the sibling, respectively, by the "Oslo Social Support Scale" (OSSS; Dalgard, 2006). The sum score ranges from 3 to 14. The higher the sum score, the stronger the social support.
Sociodemographic information of the parents | 2 minutes
  Sociodemographic information of the parents, assessed from the perspective of the parents by ad-hoc items.
Relationships between siblings (SRQ) | 3 minutes
  Sibling relationship, assessed from the perspective of the siblings (from 10 years of age) by the "Sibling Relationship Questionnaire" (Bojanowski, Riestock, Nisslein, Weschenfelder-Stachwitz, & Lehmkuhl, 2015). Each item is scored on a 5-point Likert scale
  (1 to 5).
Family relationships, family dynamics and functionality (FB-A) | 3 minutes
  Family relationships, family dynamics and functionality, assessed from the perspective of the parents, of the chronically-ill children/adolescents and from the sibling, respectively by "Familienbögen" (FB-A; Cierpka & Frevert, 1994). Items are rated on a four-point Likert scale (0 to 3)
Interpersonal problems (IIP-32) | 3 minutes
  Interpersonal problems assessed from the perspective of the parents by the "Inventory of Interpersonal Problems-32" (IIP-32; Thomas, Brähler, & Strauß, 2011). Items are rated on a four-point Likert scale from 0 (not at all) to 4 (extremely). It provides an overall score and eight subscale scores.
Familial predispositions (FaBel) | 3 minutes
  familial predispositions assessed from the perspective of the parents by the "Familien-Belastungs-Fragebogen" (FaBel; Ravens-Sieberer, 2001). Items are rated on a four-point Likert scale ranging from 1 (is not right at all) to 4 (is completely right).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Boettcher J, Hohmann S, Daubmann A, Denecke J, Muntau AC, Wiegand-Grefe S, Zapf H. The Family Stress Model in families of children with rare diseases: a cross-sectional multilevel path analysis for understanding family dynamics. Front Public Health. 2025 Nov 18;13:1713613. doi: 10.3389/fpubh.2025.1713613. eCollection 2025. PMID 41341441
- [Derived] Boettcher J, Nazarian R, Fuerboeter M, Liedtke A, Wiegand-Grefe S, Reinshagen K, Boettcher M. Mental Health of Siblings of Children with Rare Congenital Surgical Diseases during the COVID-19 Pandemic. Eur J Pediatr Surg. 2022 Oct;32(5):422-428. doi: 10.1055/s-0041-1740978. Epub 2021 Dec 31. PMID 34972234